CLINICAL TRIAL: NCT02603172
Title: A Three-part Open-label, Non-randomised, Dose-escalation Study to Investigate the Safety and Tolerability of GSK3039294 Administered as a Single Dose to Healthy Volunteers, and as Repeat Dose to Healthy Volunteers and Patients With Systemic Amyloidosis
Brief Title: A Safety Study of GSK3039294 in Healthy Volunteers and Patients With Systemic Amyloidosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A new study will be initiated in order to specifically investigate cardiac safety
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201664; 2015-003088-13 (EudraCT Number)
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: Amyloidosis
Keywords: GSK3039294; GSK2315698; systemic amyloidosis; CPHPC; dose-escalation
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part A: Cohort 1 (Experimental): Subjects will receive a single dose of GSK3039294 (Dose level 1) on Day 1 and will remain in-house until Day 4. Wash-out will take place from Day 5 to Day 14. Subjects will receive Dose level 2 on Day 15 (Period 2).
  Interventions: Drug: GSK3039294
- Part A: Cohort 2 (Experimental): Subjects will receive a single dose of GSK3039294 (Dose level 3) on Day 1 and will remain in-house until Day 4. Wash-out will take place from Day 5 to Day 14. Subjects will receive Dose level 4 on Day 15 (Period 2).
  Interventions: Drug: GSK3039294
- Part B: Cohort 3a (Experimental): Subjects will receive repeat dosing of GSK3039294 for a total of 21 days. The dose will be escalated every week throughout the study duration. Subjects will first receive a low dose given once daily. After 7 days, if well tolerated, the total daily dose will be increased and, GSK3039294 will be given, for example, as twice daily dosing for 7 days. At the end of this 7 day period and if previous dosing was well tolerated, the dose will be increased to a maximum daily dose that will not exceed pre-clinical safety exposure limits. On Day 4 and 5 GSK3039294 will be administered under fasted and fed conditions, respectively, to investigate the food effect on the PK.
  Interventions: Drug: GSK3039294
- Part B: Cohort 3b (Experimental): Subjects will be enrolled in Cohort 3b only if required for further investigation. Subjects will receive GSK3039294 for 21 consecutive days and more than one dose level or regimen may be investigated, for example on the first 10 days the dose may be administered thrice daily, and on the last 11 days may be administered twice daily.
  Interventions: Drug: GSK3039294
- Part C: Cohort 4 (Experimental): Subjects will receive repeat dosing of GSK3039294 at the predicted optimal clinical dose determined from Part B for a total of 21 days.
  Interventions: Drug: GSK3039294

INTERVENTIONS:
Drug: GSK3039294 — GSK3039294 will be provided as white, opaque capsules. A single capsule or multiple capsules (20 mg to 200 mg), depending on the dosage required, will be taken orally with water.

SUMMARY:
GSK3039294 has been developed in order to offer an orally available alternative to parenteral CPHPC (GSK2315698 [metabolite of GSK3039294]) for plasma serum amyloid P component (SAP) depletion prior to use of anti SAP monoclonal antibody (mAb) in the treatment of systemic amyloidosis. This phase 1 study is intended to study safety, tolerability and pharmacokinetic (PK) profile of GSK3039294 in humans. This study consists of three parts. Part A will evaluate safety and tolerability of single doses of GSK3039294 in healthy subjects, Part B will evaluate safety and tolerability of repeat doses of GSK3039294 in healthy subjects, and Part C will evaluate safety and tolerability of repeat doses of GSK3039294 in subjects with systemic amyloidosis. Part A is a single dose, open label, dose escalation study. Two cohorts of subjects will be enrolled to provide data from 6 subjects per cohort and up to 4 different doses (2 dose levels per cohort) of GSK3039294 will be tested. For Cohorts 1 and 2, each subject may take part in two dosing periods. Part B is repeat dose, open label, dose escalation study. Sufficient number of subjects will be enrolled in Cohort 3a to ensure 6 completers (Cohort 3b will be conducted if required) and GSK3039294 will be administered repeatedly for a total of 21 days. Each subject will take part in a single study period. In Part C a single dose level of GSK3039294 will be tested for 21 days repeat dose, in 12 subjects with systemic amyloidosis. Each subject will take part in a single study period. The total duration for Part A is approximately 8 weeks, Part B is approximately 8-9 weeks, and Part C is approximately 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 70 years of age inclusive at the time of signing the informed consent.
* Non-smokers and Smokers. Smokers (<5 /day) are permitted but must be willing to abstain for the duration of residential study sessions and / or dosing period (whichever is longer).
* Body weight >50 kilograms (kg) and body mass index (BMI) within the range 18.5-32 kg/square meter (m^2) (inclusive) and excluding the effects of peripheral oedema.
* Male or female
* Female subjects are eligible to participate if they are of non-childbearing potential defined as premenopausal females with a documented tubal ligation or hysterectomy or bilateral oophorectomy; or postmenopausal defined as 12 month of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli-international units (MIU)/milliliter (mL) and estradiol < 40 picograms (pg)/mL (147 picomoles [pmol]/liter [L]) is confirmatory
* Male subjects with female partners of child bearing potential must comply with one of the following contraception requirements from the time of first dose of study medication until completion of the follow-up visit: (a.) Vasectomy with documentation of azoospermia; (b.) Male condom plus partner use of one of the following contraceptive options: Contraceptive subdermal implant that meets the effectiveness criteria of a <1% rate of failure per year, as stated in the product label, Intrauterine device or intrauterine system that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label, Oral Contraceptive either combined or progestogen alone, Injectable progestogen, Contraceptive vaginal ring, Percutaneous contraceptive patches, Occlusive cap (female diaphragm or cervical/vault cap) with a vaginal spermicide (foam, gel, cream or suppository). These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.
* Additional Inclusion Criteria - Healthy Volunteers: Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Additional Inclusion Criteria - Healthy Volunteers: A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Additional Inclusion Criteria - Healthy Volunteers: aspartate aminotransferase (AST), alanine transaminase (ALT), alkaline phosphatase and bilirubin <=1.5 upper limit of normal (ULN) (isolated bilirubin >1.5 ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Additional Inclusion Criteria - Patients: Subject medically diagnosed with systemic amyloidosis
* Additional Inclusion Criteria - Patients: serum amyloid P component (SAP) scan identifying amyloid at any anatomical site, including subset of patients with moderate-large amyloid load in the liver
* Additional Inclusion Criteria - Patients: Up to and including New York Heart Association (NYHA) class 2 with a stable clinical cardiac status 12 weeks prior to screening
* Additional Inclusion Criteria - Patients: For Amyloid Light-chain (AL) amyloidosis patients, >=12 months post-chemotherapy with a stable free light chain (FLC) ratio in the preceding 4 months
* Additional Inclusion Criteria - Patients: estimated glomerular filtration rate (eGFR) >50 mL/minute
* Additional Inclusion Criteria - Patients: Alanine amino transferase (ALT) <=3x upper limit of normal (ULN) and bilirubin <=1.5x ULN (isolated bilirubin >1.5 xULN is acceptable if bilirubin was fractionated and direct bilirubin <35%), irrespective of alkaline phosphatase (ALP) level
* Additional Inclusion Criteria - Patients: Subject is ambulant and capable of attending the clinical unit

Exclusion Criteria:

* Prohibited medication
* History of regular alcohol consumption within 6 months of the study defined as: For United Kingdom (UK )sites - healthy volunteers: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or metabolite thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen
* A positive test for human immunodeficiency virus (HIV) antibody
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 84 days
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer). Prior to Part A for subjects participating in Parts A and B
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day Lactating females
* Poor or unsuitable venous access
* Additional Exclusion Criteria - Healthy Volunteer: Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Additional Exclusion Criteria - Healthy Volunteer: corrected QT interval using Fridericia's formula (QTcF) >450 milliseconds (msec) from a mean of triplicate readings triplicate readings taken 5 minutes apart
* Additional Exclusion Criteria - Patients: Subject with mean QTcF of >480 msec from a mean of triplicate readings
* Additional Exclusion Criteria - Patients: First degree heart block deemed to require pacing; Second degree atrioventricular (AV) block Mobitz Type II; Trifasicular block; Ventricular tachyarrthymias - with the exception of bundle branch block, atrial fibrillation & first degree heart block not requiring pacing, or second degree AV block Mobitz Type I
* Additional Exclusion Criteria - Patients: 24 hour proteinuria >=5 g
* Additional Exclusion Criteria - Patients: A syncopal episode, of any causation, within 4 weeks of screening
* Additional Exclusion Criteria - Patients: Average systolic blood pressure (SBP) <=90 millimeter of mercury (mmHg) at Screening from triplicate readings
* Additional Exclusion Criteria - Patients: Implantable cardiac defibrillator (ICD)
* Additional Exclusion Criteria - Patients: Evidence of severe cardiac dysfunction within 12 months of screening, as diagnosed by a cardiologist, using Echocardiography or cardiac magnetic resonance imaging (MRI) i.e. markedly impaired ejection fraction (EF) (EF < 50% for cardiac amyloidosis patients), or cardiac imaging parameters of severe diastolic dysfunction (grade 3 or 4)
* Additional Exclusion Criteria - Patients: Anaemia hemoglobin <9 g/deciliter (dL)
* Additional Exclusion Criteria - Patients: Uncontrolled hypertension in a known hypertensive patient, or fulfilling diagnostic criteria of essential hypertension at screening
* Additional Exclusion Criteria - Patients: Presence of any co-morbid condition (e.g. severe or unstable coronary artery disease; moderate to severe chronic obstructive pulmonary disease) which in the opinion of the investigator would increase the potential risk to the subject
* Additional Exclusion Criteria - Patients: Non-amyloidosis causes of chronic liver disease (with the exception of Gilbert's syndrome or clinically asymptomatic gallstones)
* Additional Exclusion Criteria - Patients: Diabetes Mellitus
* Additional Exclusion Criteria - Patients: Glycosuria at Screening
* Additional Exclusion Criteria - Patients: Urine power of Hydrogen (pH) <6.0 at screening
* Additional Exclusion Criteria - Patients: Hypoalbuminemia (<30 nanomoles [nmol]/L)
* Additional Exclusion Criteria - Patients: Hypophosphatemia (less than 0.8 millimoles [mmol]/L)
* Additional Exclusion Criteria - Patients: Prothombin time >1.5xULN
* Additional Exclusion Criteria - Patients: Malabsorption syndrome of any aetiology
* Additional Exclusion Criteria - Patients: Compassionate use of CPHPC (GSK2315698) or participation in a separate clinical trial involving CPHPC within 3 months of screening
* Additional Exclusion Criteria - Patients: Currently taking any of the following esterase-cleaved prodrug medications: cerebyx, aquavan, spectracef, hepsera, viread
* Additional Exclusion Criteria - Patients: Anticoagulation therapy within 4 weeks of Screening
* Additional Exclusion Criteria - Patients: Currently receiving or have received within 12 weeks of screening immunosuppressive anti-cytokine monoclonal antibodies (e.g. anti-tumor necrosis factor [anti-TNF] or anti-interleukin 1[anti-IL-1]), disease modifying drugs (e.g. methotrexate, gold or cyclophosphamide), or high-dose infusional steroids (e.g. methylprednisolone), with the exception of low-dose maintenance oral corticosteroids (e.g. <=30 milligrams (mg) prednisolone per day)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in the United Kingdom from 12-May-2016 to 10-May-2017. The study was terminated due to safety reasons during conduct of Part B (end of Cohort 3) whereas Cohort 4A and 4B were not recruited in Part B and Part C was not initiated.
Pre-assignment Details: This was 3 parts study, participants received GSK3039294: single ascending dose in Part A; repeated dose in Part B; repeat dose in systemic amyloidosis in Part C. Participants in Part A also participated in Part B of the study.
Groups:
- GSK3039294 200 mg + GSK3039294 600 mg: In Part A Cohort 1, participants received a single dose of GSK3039294 (dose level 1) 200 milligram (mg) capsules, orally, once on Day 1 and stayed in-house until Day 4; followed by washout period from Day 5 to 14; followed by a single dose of GSK3039294 (dose level 2) 600 mg capsules, orally, once on Day 1 and stayed in-house until Day 4. The remaining participants received the same dose of GSK3039294 (dose level 3) 600 mg capsules, orally, once on Day 1 in Part A Cohort 2.
- GSK3039294 200 mg + GSK3039294 600 mg/GSK3039294 600 mg QD: In Part A Cohort 1, participants received a single dose of GSK3039294 (dose level 1) 200 milligram (mg) capsules, orally, once on Day 1 and stayed in-house until Day 4; followed by washout period from Day 5 to 14; followed by a single dose of GSK3039294 (dose level 2) 600 mg capsules, orally, once on Day 1 and stayed in-house until Day 4. The remaining participants received the same dose of GSK3039294 (dose level 3) 600 mg capsules, orally, once on Day 1 in Part A Cohort 2. In Part B Cohort 3, participants received GSK3039294 600 mg capsules, orally, under fed condition, once daily (QD) for 7 days.
- GSK3039294 600 mg +GSK3039294 1200 mg: In Part A Cohort 2, participants received GSK3039294 (dose level 3) 600 mg capsules, orally, once on Day 1, and stayed in-house until Day 4; followed by washout period from Day 5 to 14; followed by a single dose of GSK3039294 (dose level 4) 1200 mg capsules, orally, once on Day 1 and stayed in-house until Day 4.
- GSK3039294 600 mg +GSK3039294 1200 mg/GSK3039294 600 mg QD: In Part A Cohort 2, participants received GSK3039294 (dose level 3) 600 mg capsules, orally, once on Day 1, and stayed in-house until Day 4; followed by washout period from Day 5 to 14; followed by a single dose of GSK3039294 (dose level 4) 1200 mg capsules, orally, once on Day 1 and stayed in-house until Day 4. In Part B Cohort 3, participants received GSK3039294 600 mg capsules, orally, under fed condition, once daily (QD) for 7 days.
- GSK3039294 600 mg QD: In Part B Cohort 3, participants received GSK3039294 600 mg capsules, orally, under fed condition, QD for 7 days.
- GSK3039294 (Cohort 4a): Participants were planned to receive repeat dose of GSK3039294 for 21 days in cohort 4a. The dose level was to be adjusted once during the 21 days. Cohort 4a was not initiated due to safety reasons during conduct of Part B (Cohort 3).
- GSK3039294 (Cohort 4b): Participants were planned to receive repeat dose of GSK3039294 for 21 days in cohort 4b. The dose level was to be adjusted once during the 21 days. Cohort 4b was not initiated due to safety reasons during conduct of Part B (Cohort 3).
- Part C: GSK3039294: Participants were planned to receive repeat dose of GSK3039294 at the predicted optimal clinical dose determined from Part B for a total of 21 days.
Period: Part A (Approximately 16 Weeks)
Arm/Group | GSK3039294 200 mg + GSK3039294 600 mg | GSK3039294 200 mg + GSK3039294 600 mg/GSK3039294 600 mg QD | GSK3039294 600 mg +GSK3039294 1200 mg | GSK3039294 600 mg +GSK3039294 1200 mg/GSK3039294 600 mg QD | GSK3039294 600 mg QD | GSK3039294 (Cohort 4a) | GSK3039294 (Cohort 4b) | Part C: GSK3039294
Started | 7 | 1 | 8 | 1 | 0 | 0 | 0 | 0
Completed | 7 | 1 | 7 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part B (Approximately 7 Weeks)
Arm/Group | GSK3039294 200 mg + GSK3039294 600 mg | GSK3039294 200 mg + GSK3039294 600 mg/GSK3039294 600 mg QD | GSK3039294 600 mg +GSK3039294 1200 mg | GSK3039294 600 mg +GSK3039294 1200 mg/GSK3039294 600 mg QD | GSK3039294 600 mg QD | GSK3039294 (Cohort 4a) | GSK3039294 (Cohort 4b) | Part C: GSK3039294
Started | 0 | 1 | 0 | 1 | 6 | 0 | 0 | 0
Completed | 0 | 1 | 0 | 1 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C (Approximately 13 Weeks)
Arm/Group | GSK3039294 200 mg + GSK3039294 600 mg | GSK3039294 200 mg + GSK3039294 600 mg/GSK3039294 600 mg QD | GSK3039294 600 mg +GSK3039294 1200 mg | GSK3039294 600 mg +GSK3039294 1200 mg/GSK3039294 600 mg QD | GSK3039294 600 mg QD | GSK3039294 (Cohort 4a) | GSK3039294 (Cohort 4b) | Part C: GSK3039294
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated due to safety reasons during conduct of Part B (end of Cohort 3) whereas Cohort 4A and 4B were not recruited in Part B and Part C was not initiated.
Groups:
- GSK3039294 200 mg + GSK3039294 600 mg: In Part A Cohort 1, participants received a single dose of GSK3039294 (dose level 1) 200 mg capsules, orally, once on Day 1 and stayed in-house until Day 4; followed by washout period from Day 5 to 14; followed by a single dose of GSK3039294 (dose level 2) 600 mg capsules, orally, once on Day 1 and stayed in-house until Day 4. The remaining participants received the same dose of GSK3039294 (dose level 3) 600 mg capsules, orally, once on Day 1 in Part A Cohort 2.
- GSK3039294 200 mg + GSK3039294 600 mg/GSK3039294 600 mg QD: In Part A Cohort 1, participants received a single dose of GSK3039294 (dose level 1) 200 mg capsules, orally, once on Day 1 and stayed in-house until Day 4; followed by washout period from Day 5 to 14; followed by a single dose of GSK3039294 (dose level 2) 600 mg capsules, orally, once on Day 1 and stayed in-house until Day 4. The remaining participants received the same dose of GSK3039294 (dose level 3) 600 mg capsules, orally, once on Day 1 in Part A Cohort 2. In Part B Cohort 3, participants received GSK3039294 600 mg capsules, orally, under fed condition, QD for 7 days.
- GSK3039294 600 mg +GSK3039294 1200 mg/GSK3039294 600 mg QD: In Part A Cohort 2, participants received GSK3039294 (dose level 3) 600 mg capsules, orally, once on Day 1, and stayed in-house until Day 4; followed by washout period from Day 5 to 14; followed by a single dose of GSK3039294 (dose level 4) 1200 mg capsules, orally, once on Day 1 and stayed in-house until Day 4. In Part B Cohort 3, participants received GSK3039294 600 mg capsules, orally, under fed condition, QD for 7 days.
- Total: Total of all reporting groups
Arm/Group | GSK3039294 200 mg + GSK3039294 600 mg | GSK3039294 200 mg + GSK3039294 600 mg/GSK3039294 600 mg QD | GSK3039294 600 mg +GSK3039294 1200 mg | GSK3039294 600 mg +GSK3039294 1200 mg/GSK3039294 600 mg QD | GSK3039294 600 mg QD | GSK3039294 (Cohort 4a) | GSK3039294 (Cohort 4b) | Part C: GSK3039294 | Total
Number analyzed (Participants) | 7 | 1 | 8 | 1 | 6 | 0 | 0 | 0 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.4 (8.48) | 26.0 (NA) — Standard Deviation could not be calculated as only one participant was analyzed | 42.1 (13.12) | 38.0 (NA) — Standard Deviation could not be calculated as only one participant was analyzed | 36.3 (7.79) |  |  |  | 38.2 (9.235)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 7 | 1 | 8 | 1 | 6 | 0 | 0 | 0 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  CENTRAL/SOUTH ASIAN HERITAGE | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  BLACK OR AFRICAN AMERICAN | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | 6 | 1 | 7 | 1 | 6 | 0 | 0 | 0 | 21

OUTCOME MEASURES:

1. Primary Outcome: Part A:Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participants or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization clinical chemor prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect and other important medical events judged by the investigator that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention. Safety population consist of all participants who received at least one dose of the study medication.
Time Frame: Up to Day 14
Population: Safety population.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: GSK3039294 200 mg: Participants received a single dose of GSK3039294 (dose level 1) 200 mg capsules, orally, once on Day 1 and stayed in-house until Day 4 in cohort 1.
- Part A: GSK3039294 600 mg: Participants received a single dose of GSK3039294 (dose level 2) 600 mg capsules, orally, once on Day 1 and stayed in-house until Day 4 in cohort 1. The remaining participants received the same dose of GSK3039294 (dose level 3) 600 mg, capsules, orally, once on Day 1 and stayed in-house until Day 4 in cohort 2. A washout period was maintained from Day 5 to 14 between two treatment cohorts.
- Part A: GSK3039294 1200 mg: Participants received a single dose of GSK3039294 (dose level 4) 1200 mg, capsules, orally, once on Day 1 and stayed in-house until Day 4 in cohort 2.
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
Participants
  Any AEs | 1 | 6 | 5
  Any SAEs | 0 | 0 | 0

2. Primary Outcome: Part A: Number of Participants With Emergent Clinical Chemistry by Potentially Clinical Importance (PCI) Criteria
Description: PCI ranges for the clinical chemistry parameters were as follows : albumin (low: <0.86 gram [g] per liter [L]), calcium (low: <0.91 millimole [mmol]/L and high: >1.06 mmol/L), glucose (low: <0.71 mmol/L and high: >1.41 mmol/L), magnesium (low: <0.63 mmol/L and high: >1.03 mmol/L), phosphorous (low: <0.80 mmol/L and high: >1.14 mmol/L), potassium (low: <0.86 mmol/L and high: >1.10 mmol/L), sodium (low: <0.96 mmol/L and high: >1.03 mmol/L), and total carbon dioxide (CO2) (low: <0.86 mmol/L and high: >1.14 mmol/L).
Time Frame: Day 1
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
Participants
  Albumin: low | 0 | 0 | 0
  Albumin: high | 0 | 0 | 0
  Calcium: low | 0 | 0 | 0
  Calcium: high | 0 | 0 | 0
  Glucose: low | 0 | 0 | 0
  Glucose: high | 0 | 0 | 0
  Potassium: low | 0 | 0 | 0
  Potassium: high | 0 | 0 | 0
  Sodium: low | 0 | 0 | 0
  Sodium: high | 0 | 0 | 0

3. Primary Outcome: Part A: Number of Participants With Emergent Hematology by PCI Criteria
Description: PCI ranges for the hematology parameters were as follows: white blood cell (WBC) count (low: <0.67 10^9 cells/L and high: >1.82 10^9 cells/L), neutrophil count (low: <0.83 10^9 cells/L), hemoglobin (high: >1.03 g/L in male, >1.13 g/L in female), hemocrit (high: >1.02 proportion of red blood cell [RBC] in blood for male, >1.17 proportion of RBC in blood for female), platelet count (low: <0.67 10^9 cells/L and high: 1.57 10^9 cells/L), and lymphocytes (low: <0.81 10^9 cells/L).
Time Frame: Day 1
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
Participants
  Hematocrit: low | 0 | 0 | 0
  Hematocrit: high | 0 | 0 | 0
  Hemoglobin: low | 0 | 0 | 0
  Hemoglobin: high | 0 | 0 | 0
  Leukocytes: low | 0 | 0 | 0
  Leukocytes: high | 0 | 0 | 0
  Lymphocytes: low | 0 | 0 | 0
  Lymphocytes: high | 0 | 0 | 0
  Neutrophils: low | 0 | 0 | 0
  Neutrophils: high | 0 | 0 | 0

4. Primary Outcome: Part A: Number of Participants With Abnormal Urinalysis Data by Dipstick
Description: Urine samples were collected and urinalysis included analysis of specific gravity, potential of hydrogen (pH), glucose, protein, blood, ketones by dipstick. The dipstick test gives results in a semi-quantitative manner.
Time Frame: Day 1
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
Participants | 0 | 0 | 0

5. Primary Outcome: Part A: Mean Change From Baseline in 12-lead Electrocardiogram (ECG)
Description: Triplicate ECG was measured in semi-supine position after 5 minutes (min) rest. A single 12-lead ECG was measured by using ECG machine that automatically measured PR, QRS, QT, and Fridericia's formula (QTcF) intervals. Baseline is defined as the latest available assessment pre the first dose of study drug within each period in Part A. Change from Baseline was calculated as any visit post Baseline value minus Baseline value.
Time Frame: Baseline (pre-dose) and 15, 30 minutes, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
Millisecond
  PR interval: 15 minutes | 0.5 (5.47) | 0.9 (7.05) | -0.3 (3.47)
  PR interval: 30 minutes | -0.3 (6.24) | 3.1 (5.65) | 0.2 (5.35)
  PR interval: 1 hour | -2.3 (8.72) | 3.2 (6.06) | 0.3 (7.19)
  PR interval: 2 hour | -0.3 (4.82) | 0.2 (5.50) | 0.3 (5.42)
  PR interval: 4 hour | -8.3 (6.41) | -7.3 (8.22) | -7.1 (4.66)
  PR interval: 6 hour | -6.8 (7.04) | -7.6 (9.60) | -4.0 (6.98)
  PR interval: 8 hour | -5.0 (6.48) | -6.1 (8.38) | -5.0 (5.27)
  PR interval: 12 hour | -3.8 (7.42) | -6.1 (7.77) | -4.7 (9.69)
  PR interval: 24 hour | -0.3 (8.72) | -2.8 (9.23) | -1.5 (6.51)
  PR interval: 48 hour | 4.2 (10.75) | 0.9 (8.67) | 1.0 (4.44)
  PR interval: 72 hour | -3.9 (12.95) | -1.7 (11.80) | -5.3 (5.43)
  QRS duration: 15 minutes | -0.0 (2.28) | 0.9 (3.76) | -1.3 (2.25)
  QRS duration: 30 minutes | 0.7 (1.89) | 0.9 (2.70) | -0.3 (1.63)
  QRS duration: 1 hour | 0.3 (3.49) | 0.1 (2.61) | -0.1 (1.69)
  QRS duration: 2 hour | -0.3 (2.28) | 0.1 (1.85) | -0.6 (3.55)
  QRS duration: 4 hour | 0.8 (4.12) | 1.0 (3.83) | 1.5 (3.32)
  QRS duration: 6 hour | -0.6 (2.65) | -0.4 (2.59) | -1.2 (2.64)
  QRS duration: 8 hour | -0.0 (2.71) | 0.4 (3.26) | -0.6 (3.05)
  QRS duration: 12 hour | 0.7 (2.05) | 1.0 (4.28) | 0.9 (3.85)
  QRS duration: 24 hour | -0.2 (1.70) | 0.1 (2.40) | -0.5 (2.82)
  QRS duration: 48 hour | 1.3 (2.57) | 2.0 (4.18) | 0.3 (3.79)
  QRS duration: 72 hour | 0.5 (1.84) | 2.7 (3.39) | -2.0 (4.83)
  QT interval: 15 minutes | 5.6 (6.72) | -2.4 (13.95) | -3.0 (5.51)
  QT interval: 30 minutes | 1.3 (7.81) | 0.4 (10.44) | -2.5 (5.31)
  QT interval: 1 hour | 4.8 (11.90) | 3.0 (12.77) | -3.8 (8.45)
  QT interval: 2 hour | 3.2 (7.12) | 2.4 (9.32) | -1.3 (5.20)
  QT interval: 4 hour | -19.5 (4.83) | -22.5 (10.73) | -18.7 (11.62)
  QT interval: 6 hour | -17.8 (8.76) | -19.2 (12.40) | -21.0 (15.15)
  QT interval: 8 hour | -11.0 (17.22) | -15.8 (10.78) | -14.2 (12.45)
  QT interval: 12 hour | -6.2 (10.62) | -13.1 (13.87) | -16.8 (11.77)
  QT interval: 24 hour | -3.7 (12.56) | -9.5 (8.32) | -4.5 (8.43)
  QT interval: 48 hour | -8.0 (16.27) | -16.4 (10.05) | -19.3 (23.78)
  QT interval: 72 hour | -26.0 (23.84) | -29.6 (14.29) | -27.5 (16.36)
  QTcF interval: 15 minutes | -0.7 (2.58) | 1.1 (9.02) | -1.5 (6.95)
  QTcF interval: 30 minutes | -3.6 (4.56) | 2.0 (7.54) | -0.2 (6.75)
  QTcF interval: 1 hour | -0.6 (4.07) | 1.4 (6.37) | 0.7 (6.35)
  QTcF interval: 2 hour | 0.3 (6.54) | 0.0 (7.53) | 1.1 (4.99)
  QTcF interval: 4 hour | -2.6 (8.50) | -0.3 (10.31) | 1.6 (8.98)
  QTcF interval: 6 hour | -5.6 (5.98) | -5.2 (8.96) | -2.9 (11.44)
  QTcF interval: 8 hour | -6.7 (7.28) | -5.9 (7.71) | -1.7 (8.63)
  QTcF interval: 12 hour | -3.6 (7.30) | -4.0 (8.64) | -1.4 (9.23)
  QTcF interval: 24 hour | -5.6 (7.00) | -3.0 (5.35) | -3.4 (7.88)
  QTcF interval: 48 hour | -8.3 (5.56) | -5.9 (8.39) | -1.8 (14.81)
  QTcF interval: 72 hour | -10.4 (10.32) | -9.6 (10.65) | -3.7 (13.01)

6. Primary Outcome: Part A: Mean Change From Baseline in Heart Rate by 12-lead ECG
Description: Triplicate ECG was measured in semi-supine position after 5 min rest. A single 12-lead ECG was measured by using ECG machine that automatically measures the heart rate. Baseline is defined as the latest available assessment pre the first dose of study drug within each period in Part A. Change from Baseline was calculated as any visit post Baseline value minus Baseline value.
Time Frame: Baseline (pre-dose) and 15, 30 minutes, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
Beats per minute
  15 minutes | -2.1 (2.90) | 0.9 (4.27) | 0.6 (1.96)
  30 minutes | -2.0 (3.10) | 0.9 (4.64) | 1.0 (2.62)
  1 hour | -2.0 (4.95) | -0.4 (3.72) | 1.8 (1.77)
  2 hour | -1.1 (3.97) | -0.7 (3.38) | 1.0 (2.27)
  4 hour | 8.1 (4.13) | 9.7 (4.29) | 8.3 (5.27)
  6 hour | 5.8 (4.21) | 5.7 (4.63) | 7.3 (3.52)
  8 hour | 2.4 (6.67) | 4.1 (4.79) | 5.2 (5.55)
  12 hour | 1.1 (2.17) | 3.8 (4.15) | 6.3 (2.69)
  24 hour | -1.2 (4.02) | 2.7 (3.33) | 0.4 (2.08)
  48 hour | -0.4 (6.70) | 4.3 (5.74) | 7.8 (8.60)
  72 hour | 6.9 (6.33) | 8.8 (6.74) | 10.8 (8.77)

7. Primary Outcome: Part A: Mean Change From Baseline in Blood Pressure (BP)
Description: Systolic BP and diastolic BP were measured in semi-supine position after 5 min rest for the participants at indicated time points. Baseline is defined as the latest available assessment pre the first dose of study drug within each period in Part A. Change from Baseline was calculated as any visit post Baseline value minus Baseline value.
Time Frame: Baseline (pre-dose) and 15, 30 minutes, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
Millimeter of mercury
  Diastolic BP: 15 minutes | -0.6 (3.11) | -0.4 (3.86) | 3.5 (4.86)
  Diastolic BP: 30 minutes | -0.1 (1.54) | 0.1 (3.72) | 2.9 (4.04)
  Diastolic BP: 1 hour | -2.0 (4.13) | -1.1 (3.53) | 0.9 (4.25)
  Diastolic BP: 2 hour | -3.1 (3.16) | -1.7 (4.95) | 1.4 (4.06)
  Diastolic BP: 4 hour | -7.3 (2.45) | -6.5 (5.83) | -2.5 (6.54)
  Diastolic BP: 6 hour | -4.7 (3.82) | -4.8 (4.80) | -0.3 (4.38)
  Diastolic BP: 8 hour | -2.0 (5.47) | -1.9 (6.16) | 0.8 (6.09)
  Diastolic BP: 12 hour | -7.1 (2.88) | -4.6 (5.77) | -2.6 (7.39)
  Diastolic BP: 24 hour | -1.6 (4.48) | -2.6 (5.52) | 2.5 (4.25)
  Diastolic BP: 48 hour | -3.0 (2.69) | -2.1 (6.35) | 0.0 (6.24)
  Diastolic BP: 72 hour | -4.7 (3.82) | -3.2 (5.54) | -0.0 (3.99)
  Systolic BP: 15 minutes | -2.0 (5.08) | 0.8 (4.74) | 1.0 (4.12)
  Systolic BP: 30 minutes | -0.7 (4.46) | -0.8 (4.59) | 1.7 (1.86)
  Systolic BP: 1 hour | -1.2 (5.79) | 0.2 (3.85) | 0.7 (2.40)
  Systolic BP: 2 hour | -2.6 (5.38) | 0.7 (5.77) | 1.8 (4.87)
  Systolic BP: 4 hour | -3.9 (5.84) | 0.1 (6.65) | 3.6 (7.27)
  Systolic BP: 6 hour | -2.3 (6.62) | -1.1 (5.91) | 1.2 (6.09)
  Systolic BP: 8 hour | -2.0 (9.37) | 1.5 (8.50) | 3.8 (7.62)
  Systolic BP: 12 hour | -3.2 (5.70) | 0.1 (7.54) | 3.6 (7.72)
  Systolic BP: 24 hour | -2.8 (5.06) | 0.1 (5.64) | 4.3 (6.75)
  Systolic BP: 48 hour | -2.2 (4.83) | 0.5 (4.88) | 3.3 (7.55)
  Systolic BP: 72 hour | -1.1 (7.84) | 3.4 (6.58) | 6.0 (5.42)

8. Primary Outcome: Part A: Mean Change From Baseline in Pulse Rate
Description: Pulse rate was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Baseline is defined as the latest available assessment pre the first dose of study drug within each period in Part A. Change from Baseline was calculated as any visit post Baseline value minus Baseline value.
Time Frame: Baseline (pre-dose) and 15, 30 minutes, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
Beats per minute
  15 minutes | 0.2 (2.15) | -0.4 (2.25) | 0.4 (3.14)
  30 minutes | -0.4 (3.06) | 0.5 (2.17) | 1.7 (2.91)
  1 hour | -0.2 (5.17) | 0.4 (3.10) | 1.3 (3.51)
  2 hour | -0.7 (1.76) | -0.3 (5.00) | 1.5 (2.36)
  4 hour | 9.3 (4.64) | 9.0 (4.90) | 7.9 (4.01)
  6 hour | 7.1 (6.71) | 4.6 (4.44) | 7.5 (3.59)
  8 hour | 4.4 (6.29) | 4.4 (5.72) | 5.0 (5.61)
  12 hour | 2.3 (3.58) | 3.8 (3.82) | 5.5 (4.01)
  24 hour | 2.1 (3.93) | 2.1 (3.22) | 1.1 (3.15)
  48 hour | 2.5 (5.53) | 4.9 (5.77) | 7.9 (9.99)
  72 hour | 9.9 (7.06) | 9.8 (7.47) | 11.1 (8.94)

9. Primary Outcome: Part A: Mean Change From Baseline in Temperature
Description: Temperature was measured in semi-supine position after 5 min rest for the participants at indicated time points. Baseline is defined as the latest available assessment pre the first dose of study drug within each period in Part A. Change from Baseline was calculated as any visit post Baseline value minus Baseline value.
Time Frame: Baseline (pre-dose) and 15, 30 minutes, 1, 2, 4, 6, 8, 12, 24, 48 and 72 hours post-dose
Population: Safety population.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
Celsius
  15 minutes | -0.18 (0.292) | -0.00 (0.339) | 0.10 (0.239)
  30 minutes | -0.14 (0.374) | -0.02 (0.369) | 0.09 (0.253)
  1 hour | -0.26 (0.469) | 0.09 (0.380) | 0.17 (0.255)
  2 hour | -0.06 (0.288) | 0.09 (0.278) | 0.21 (0.230)
  4 hour | 0.24 (0.329) | 0.27 (0.453) | 0.34 (0.350)
  6 hour | 0.24 (0.250) | 0.53 (0.318) | 0.45 (0.334)
  8 hour | -0.00 (0.438) | 0.37 (0.427) | 0.47 (0.381)
  12 hour | 0.10 (0.463) | 0.19 (0.486) | 0.36 (0.534)
  24 hour | 0.09 (0.439) | 0.12 (0.276) | 0.08 (0.271)
  48 hour | 0.05 (0.417) | 0.13 (0.334) | 0.35 (0.233)
  72 hour | 0.17 (0.413) | 0.20 (0.310) | 0.43 (0.282)

10. Primary Outcome: Part B:Number of Participants With AEs and SAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect and other important medical events judged by the investigator that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention.
Time Frame: Cohort 3: Up to Day 21; Cohort 4: Up to Day 35
Population: Safety population. Data was not collected as study was terminated, due to safety reasons during conduct of Part B (end of Cohort 3) whereas Cohort 4a and 4b were not recruited in Part B.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Cohort 3- GSK3039294 600 mg QD: Participants received GSK3039294 600 mg, capsules, orally, under fed condition, QD for 7 days in cohort 3.
- Part B: Cohort 4a- GSK3039294: Participants were planned to receive repeat dose of GSK3039294 for 21 days in cohort 4a. The dose level was to be adjusted once during the 21 days. Cohort 4a was not initiated due to safety reasons during conduct of Part B (Cohort 3).
- Part B: Cohort 4b- GSK3039294: Participants were planned to receive repeat dose of GSK3039294 for 21 days in cohort 4b. The dose level was to be adjusted once during the 21 days. Cohort 4b was not initiated due to safety reasons during conduct of Part B (Cohort 3).
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
Participants
  Any AE | 7 |  |
  Any SAE | 1 |  |

11. Primary Outcome: Part B: Number of Participants With Emergent Clinical Chemistry by PCI Criteria
Description: PCI ranges for the clinical chemistry parameters were as follows: albumin (low: <0.86 g/L), calcium (low: <0.91 mmol/L and high: >1.06 mmol/L), glucose (low: <0.71 mmol/L and high: >1.41 mmol/L), magnesium (low: <0.63 mmol/L and high: >1.03 mmol/L), phosphorous (low: <0.80 mmol/L and high: >1.14 mmol/L), potassium (low: <0.86 mmol/L and high: >1.10 mmol/L), sodium (low: <0.96 mmol/L and high: >1.03 mmol/L), and total CO2 (low: <0.86 mmol/L and high: >1.14 mmol/L).
Time Frame: Cohort 3 and 4: Up to Day 3
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
Participants
  Albumin: low | 0 |  |
  Albumin: high | 0 |  |
  Calcium: low | 0 |  |
  Calcium: high | 0 |  |
  Glucose: low | 0 |  |
  Glucose: high | 0 |  |
  Potassium: low | 0 |  |
  Potassium: high | 0 |  |
  Sodium: low | 0 |  |
  Sodium: high | 0 |  |

12. Primary Outcome: Part B: Number of Participants With Emergent Hematology by PCI Criteria
Description: PCI ranges for the hematology parameters were as follows: WBC count (low: <0.67 10^9 cells/L and high: >1.82 10^9 cells/L), neutrophil count (low: <0.83 10^9 cells/L), hemoglobin (high: >1.03 g/L in male, >1.13 g/L in female), hemocrit (high: >1.02 proportion of RBC in blood for male, >1.17 proportion of RBC in blood for female), platelet count (low: <0.67 10^9 cells/L and high: 1.57 10^9 cells/L), and lymphocytes (low: <0.81 10^9 cells/L).
Time Frame: Cohort 3 and 4: Up to Day 3
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
Participants
  Hematocrit: low | 0 |  |
  Hematocrit: high | 0 |  |
  Hemoglobin: low | 0 |  |
  Hemoglobin: high | 0 |  |
  Leukocytes: low | 0 |  |
  Leukocytes: high | 0 |  |
  Lymphocytes: low | 0 |  |
  Lymphocytes: high | 0 |  |
  Neutrophils: low | 1 |  |
  Neutrophils: high | 0 |  |

13. Primary Outcome: Part B: Number of Participants With Abnormal Urinalysis Data by Dipstick
Description: Urine samples were collected and urinalysis included analysis of specific gravity, pH, glucose, protein, blood, ketones by dipstick. The dipstick test gives results in a semi-quantitative manner.
Time Frame: Cohort 3 and 4: Up to Day 3
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
Participants | 0 |  |

14. Primary Outcome: Part B: Mean Change From Baseline in 12-lead ECG
Description: Triplicate ECG was measured in semi-supine position after 5 minutes rest. A single 12-lead ECG was measured by using ECG machine that automatically measured PR, QRS, QT, and QTcF intervals. Baseline is defined as the latest available assessment pre the first dose of study drug in Part B. Change from Baseline was calculated as any visit post Baseline value minus Baseline value.
Time Frame: Cohort 3: Baseline (pre-dose), Day 1 (1 hour), Days 2, 3, 4, 5, 6, 7 (pre-dose and 1 hour), 8 and 21; Cohort 4: Up to Day 35
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
Millisecond
  PR interval- Day 1: 1 hour | 3.4 (2.42) |  |
  PR interval- Day 2: pre-dose | 2.8 (10.57) |  |
  PR interval- Day 2: 1 hour | 5.3 (7.73) |  |
  PR interval- Day 3: pre-dose | 5.0 (8.05) |  |
  PR interval- Day 3: 1 hour | 6.1 (2.96) |  |
  PR interval- Day 4: pre-dose | 2.9 (8.21) |  |
  PR interval- Day 4: 1 hour | 6.5 (4.48) |  |
  PR interval- Day 5: pre-dose | 4.5 (6.17) |  |
  PR interval- Day 5: 1 hour | 2.9 (9.50) |  |
  PR interval- Day 6: pre-dose | 4.0 (7.57) |  |
  PR interval- Day 6: 1 hour | 6.8 (6.96) |  |
  PR interval- Day 7: pre-dose | 4.6 (7.26) |  |
  PR interval- Day 7: 1 hour | 6.1 (7.13) |  |
  PR interval- Day 8 | 7.3 (7.34) |  |
  PR interval- Day 21 | 2.5 (8.38) |  |
  QRS duration- Day 1: 1 hour | -0.1 (1.78) |  |
  QRS duration- Day 2: pre-dose | -1.3 (4.22) |  |
  QRS duration- Day 2: 1 hour | -1.3 (5.95) |  |
  QRS duration- Day 3: pre-dose | -1.5 (3.29) |  |
  QRS duration- Day 3: 1 hour | -0.2 (3.42) |  |
  QRS duration- Day 4: pre-dose | 1.8 (13.09) |  |
  QRS duration- Day 4: 1 hour | -1.1 (4.20) |  |
  QRS duration- Day 5: pre-dose | -1.4 (5.20) |  |
  QRS duration- Day 5: 1 hour | 0.6 (2.97) |  |
  QRS duration- Day 6: pre-dose | -1.2 (3.41) |  |
  QRS duration- Day 6: 1 hour | -0.5 (3.08) |  |
  QRS duration- Day 7: pre-dose | -1.5 (5.25) |  |
  QRS duration- Day 7: 1 hour | 1.1 (4.22) |  |
  QRS duration- Day 8 | -0.9 (5.61) |  |
  QRS duration- Day 21 | -1.5 (6.16) |  |
  QT interval- Day 1: 1 hour | 6.0 (7.47) |  |
  QT interval- Day 2: pre-dose | 5.9 (7.44) |  |
  QT interval- Day 2: 1 hour | 7.2 (7.44) |  |
  QT interval- Day 3: pre-dose | 1.5 (8.11) |  |
  QT interval- Day 3: 1 hour | 1.0 (12.78) |  |
  QT interval- Day 4: pre-dose | 2.9 (9.68) |  |
  QT interval- Day 4: 1 hour | 0.4 (10.60) |  |
  QT interval- Day 5: pre-dose | 1.2 (7.30) |  |
  QT interval- Day 5: 1 hour | 16.6 (16.04) |  |
  QT interval- Day 6: pre-dose | 7.7 (8.64) |  |
  QT interval- Day 6: 1 hour | 2.0 (6.12) |  |
  QT interval- Day 7: pre-dose | 2.6 (11.46) |  |
  QT interval- Day 7: 1 hour | 2.5 (12.02) |  |
  QT interval- Day 8 | 1.7 (8.21) |  |
  QT interval- Day 21 | 1.4 (12.59) |  |
  QTcF interval- Day 1: 1 hour | 1.1 (5.77) |  |
  QTcF interval- Day 2: pre-dose | 4.3 (5.00) |  |
  QTcF interval- Day 2: 1 hour | 2.7 (4.13) |  |
  QTcF interval- Day 3: pre-dose | 0.5 (3.80) |  |
  QTcF interval- Day 3: 1 hour | 0.1 (5.71) |  |
  QTcF interval- Day 4: pre-dose | -1.3 (5.49) |  |
  QTcF interval- Day 4: 1 hour | -3.8 (4.73) |  |
  QTcF interval- Day 5: pre-dose | -0.4 (5.82) |  |
  QTcF interval- Day 5: 1 hour | 2.3 (10.37) |  |
  QTcF interval- Day 6: pre-dose | -2.6 (6.92) |  |
  QTcF interval- Day 6: 1 hour | -1.0 (6.76) |  |
  QTcF interval- Day 7: pre-dose | 2.4 (5.12) |  |
  QTcF interval- Day 7: 1 hour | 0.9 (3.49) |  |
  QTcF interval- Day 8 | 0.7 (6.70) |  |
  QTcF interval- Day 21 | 7.1 (6.59) |  |

15. Primary Outcome: Part B: Mean Change From Baseline in Heart Rate by 12-lead ECG
Description: Triplicate ECG was measured in semi-supine position after 5 min rest. A single 12-lead ECG was measured by using ECG machine that automatically measures heart rate. Baseline is defined as the latest available assessment pre the first dose of study drug within each period in Part B. Change from Baseline was calculated as any visit post Baseline value minus Baseline value.
Time Frame: as for outcome 14
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
Beats per minute
  Day 1: 1 hour | -1.9 (3.92) |  |
  Day 2: pre-dose | -0.6 (4.27) |  |
  Day 2: 1 hour | -2.1 (3.94) |  |
  Day 3: pre-dose | 1.3 (4.84) |  |
  Day 3: 1 hour | -0.4 (4.72) |  |
  Day 4: pre-dose | 0.9 (4.20) |  |
  Day 4: 1 hour | -1.7 (3.65) |  |
  Day 5: pre-dose | -0.6 (3.97) |  |
  Day 5: 1 hour | 9.9 (6.62) |  |
  Day 6: pre-dose | 2.4 (4.59) |  |
  Day 6: 1 hour | -1.0 (4.78) |  |
  Day 7: pre-dose | -0.0 (5.14) |  |
  Day 7: 1 hour | -0.6 (5.92) |  |
  Day 8 | 1.5 (5.24) |  |
  Day 21 | 3.4 (8.59) |  |

16. Primary Outcome: Part B: Number of Participants With Abnormal Cardiac Telemetry Findings
Description: The cardiac monitoring was measured by using an appropriate nonimplantable recording device which is acceptable to the participants. This was evaluated the arrhythmic background of eligible cardiac amyloidosis participants such that false positive attribution of arrhythmias to GSK3039294 during repeat dosing was minimized.
Time Frame: Cohort 3: Up to Day 8
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD
Number analyzed (Participants) | 8
Participants | 1

17. Primary Outcome: Part C: Number of Participants With AEs and SAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect and other important medical events judged by the investigator that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention. This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: Up to Day 63
Population: Safety Population. Data was not collected as study was terminated due to safety reasons during conduct of Part B (end of Cohort 3) whereas Part C was not initiated.
Groups:
- Part C: GSK3039294: Participants were planned to receive repeat dosing of GSK3039294 at the predicted optimal clinical dose determined from Part B for a total of 21 days.
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

18. Primary Outcome: Part C: Number of Participants With Emergent Clinical Chemistry by PCI Criteria
Description: PCI parameters for the clinical chemistry that were planned for analysis are as follows: albumin, calcium, glucose, magnesium, phosphorous , potassium , sodium , and total CO2. This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: Up to Day 63
Population: as for outcome 17
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

19. Primary Outcome: Part C: Number of Participants With Emergent Hematology Parameters by PCI Criteria
Description: Hematology parameters that were planned for analysis were as follows: WBC count , neutrophil count , hemoglobin , hemocrit , platelet count , and lymphocytes. This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: Up to Day 63
Population: as for outcome 17
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

20. Primary Outcome: Part C: Number of Participants With Emergent Urinalysis Parameters by PCI Criteria
Description: Urine samples were planned to be collected and urinalysis included analysis of specific gravity, pH, glucose, protein, blood, ketones by dipstick. This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: Up to Day 63
Population: as for outcome 17
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

21. Primary Outcome: Part C: Number of Participants With Abnormal 12-lead ECG Findings
Description: Triplicate ECG was planned to be measured in semi-supine position after 5 minutes rest. A single 12-lead ECG was measured by using ECG machine that automatically measured PR, QRS, QT, and QTcF intervals. Baseline is defined as the latest available assessment pre the first dose of study drug within each period in Part C. Change from Baseline was calculated as any visit post Baseline value minus Baseline value. This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: Up to Day 35
Population: as for outcome 17
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

22. Primary Outcome: Part C: Number of Participants With Abnormal Vital Signs
Description: Vital signs included systolic and diastolic BP, pulse rate, heart rate and temperature. This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: Up to Day 35
Population: as for outcome 17
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

23. Primary Outcome: Part C: Number of Participants With Abnormal Cardiac Telemetry Findings
Description: The cardiac monitoring was planned to be measured by using an appropriate nonimplantable recording device which is acceptable to the participants. This was evaluated the arrhythmic background of eligible cardiac amyloidosis participants such that false positive attribution of arrhythmias to GSK3039294 during repeat dosing was minimized. This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: Up to Day 35
Population: as for outcome 17
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

24. Secondary Outcome: Part A: Area Under the Concentration-time Curve Extrapolated to Infinity (AUC[0-inf]) of GSK3039294 and GSK2315698
Description: Blood samples were collected at specified time points for GSK3039294 and GSK2315698. AUC(0-inf) was determined using standard non-compartmental methods. Pharmacokinetic (PK) population consists of all participants administered at least one dose of study medication and who had at least one PK sample taken and analyzed.
Time Frame: Pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 and 48 hours post-dose
Population: PK population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
Hour*nanogram per milliliter (h*ng/mL)
  GSK3039294: n= 0, 0, 0: number analyzed (Participants) | 0 | 0 | 0
  GSK2315698: n= 8, 16, 8 | 7980.0 (28.17) | 23432.6 (23.43) | 41502.4 (14.75)

25. Secondary Outcome: Part A: AUC(0-inf) Corrected for Dose of Prodrug (AUC[0-inf]/D) of GSK3039294 and GSK2315698
Description: Blood samples were collected at specified time points for GSK3039294 and GSK2315698. AUC(0-inf)/D was determined using standard non-compartmental methods.
Time Frame: Pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 and 48 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
h*ng/mL/mg
  GSK3039294: n= 0, 0, 0: number analyzed (Participants) | 0 | 0 | 0
  GSK2315698: n= 8, 16, 8 | 39.90 (28.17) | 39.05 (23.43) | 34.59 (14.75)

26. Secondary Outcome: Part A: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-t]) of GSK3039294 and GSK2315698
Description: Blood samples were collected at specified time points for GSK3039294 and GSK2315698. AUC(0-t) was determined using standard non-compartmental methods.
Time Frame: Pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 and 48 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
h*ng/mL
  GSK3039294: n= 0, 9, 4: number analyzed (Participants) | 0 | 9 | 4
  GSK3039294: n= 0, 9, 4 |  | 10.03 (47.06) | 18.76 (30.31)
  GSK2315698: n= 8, 16, 8 | 7751.0 (29.19) | 23276.5 (23.61) | 41261.4 (14.75)

27. Secondary Outcome: Part A: AUC(0-t) Corrected for Dose of Prodrug (AUC[0-t]/D) of GSK3039294 and GSK2315698
Description: Blood samples were collected at specified time points for GSK3039294 and GSK2315698. AUC(0-t)/D was determined using standard non-compartmental methods.
Time Frame: Pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 and 48 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
h*ng/mL/mg
  GSK3039294: n= 0, 9, 4: number analyzed (Participants) | 0 | 9 | 4
  GSK3039294: n= 0, 9, 4 |  | 0.017 (47.06) | 0.016 (30.31)
  GSK2315698: n= 8, 16, 8 | 38.75 (29.19) | 38.79 (23.61) | 34.38 (14.75)

28. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of GSK3039294 and GSK2315698
Description: Blood samples were collected at specified time points for GSK3039294 and GSK2315698. Cmax was determined using standard non-compartmental methods.
Time Frame: Pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 and 48 hours post-dose
Population: PK population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). NA indicates that data could not be calculated because only one participant was analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
ng/mL
  GSK3039294: n= 1, 10, 6: number analyzed (Participants) | 1 | 10 | 6
  GSK3039294: n= 1, 10, 6 | 30.60 (NA) — NA indicates that data could not be calculated because only one participant was analyzed. | 14.82 (18.06) | 23.62 (56.24)
  GSK2315698: n= 8, 16, 8 | 3.581 (23.84) | 3.058 (21.78) | 2.476 (9.10)

29. Secondary Outcome: Part A: Cmax Corrected for Dose of Prodrug (Cmax/D) of GSK3039294 and GSK2315698
Description: Blood samples were collected at specified time points for GSK3039294 and GSK2315698. Cmax/D was determined using standard non-compartmental methods.
Time Frame: Pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 and 48 hours post-dose
Population: PK population. Data could not be calculated because only one participant was analyzed. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). NA indicates that data could not be calculated because only one participant was analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
ng/mL/mg
  GSK3039294: n= 1, 10, 6: number analyzed (Participants) | 1 | 10 | 6
  GSK3039294: n= 1, 10, 6 | 0.153 (NA) — NA indicates that data could not be calculated because only one participant was analyzed. | 0.025 (18.06) | 0.020 (56.24)
  GSK2315698: n= 8, 16, 8 | 3.581 (23.84) | 3.058 (21.78) | 2.476 (9.10)

30. Secondary Outcome: Part A: Terminal Half-life (t1/2) of GSK3039294 and GSK2315698
Description: Blood samples were collected at specified time points for GSK3039294 and GSK2315698. t1/2 was determined using standard non-compartmental methods.
Time Frame: Pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 and 48 hours post-dose
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
Hours
  GSK3039294: n= 0, 0, 0: number analyzed (Participants) | 0 | 0 | 0
  GSK2315698: n= 8, 16, 8 | 5.097 (29.60) | 6.093 (7.43) | 5.907 (7.12)

31. Secondary Outcome: Part A: Time to Reach Cmax (Tmax) of GSK3039294 and GSK2315698
Description: Blood samples were collected at specified time points for GSK3039294 and GSK2315698. tmax was determined using standard non-compartmental methods.
Time Frame: Pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24 and 48 hours post-dose
Population: as for outcome 24
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg
Number analyzed (Participants) | 8 | 16 | 8
Hours
  GSK3039294: n= 1, 10, 6: number analyzed (Participants) | 1 | 10 | 6
  GSK3039294: n= 1, 10, 6 | 0.750 [0.75 to 0.75] | 0.500 [0.25 to 1.50] | 0.867 [0.25 to 1.52]
  GSK2315698: n= 8, 16, 8 | 5.000 [3.02 to 5.12] | 6.000 [4.00 to 8.27] | 6.000 [1.580 to 8.00]

32. Secondary Outcome: Part B: Area Under the Concentration-time Curve From Time Zero to 6 Hours Post Dose (AUC[0-6]) of GSK3039294 and GSK2315698
Description: Blood samples were collected at specified time points for GSK3039294 and GSK2315698. AUC(0-6) was determined using standard non-compartmental methods.
Time Frame: Cohort 3- Day 4 and 5: pre-dose, and 0.5, 1, 2, 3, 4, and 6 hours post-dose; Cohort 4: Day 4 (pre-dose), Day 5 (pre-dose and 0.5, 1, 2, 3, 4, and 6 hours post-dose)
Population: PK population. Data was not collected as study was terminated, due to safety reasons during conduct of Part B (end of Cohort 3) whereas Cohort 4a and 4b were not recruited in Part B. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
h*ng/mL
  GSK3039294: Day 4 (n= 0, 0, 0): number analyzed (Participants) | 0 | 0 | 0
  GSK2315698: Day 4 (n= 6, 0, 0): number analyzed (Participants) | 6 | 0 | 0
  GSK2315698: Day 4 (n= 6, 0, 0) | 6899.8 (19.72) |  |
  GSK3039294: Day 5 (n= 0, 0, 0): number analyzed (Participants) | 0 | 0 | 0
  GSK2315698: Day 5 (n= 8, 0, 0) | 8900.1 (35.27) |  |

33. Secondary Outcome: Part B: AUC(0-inf) of GSK3039294 and GSK2315698
Description: Blood samples were collected at specified time points for GSK3039294 and GSK2315698. AUC(0-inf) was determined using standard non-compartmental methods.
Time Frame: as for outcome 32
Population: PK population. Data was not collected for Cohort 4a and 4b as study was terminated due to safety reasons during conduct of Part B (end of Cohort 3). Data was not calculated for Cohort 3 as the concentration-time data does not provide an accurate representation of the terminal elimination phase for the drug. Hence, AUC (0-inf) was not derived.
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 0 | 0 | 0

34. Secondary Outcome: Part B: AUC([0-inf]/D) of GSK3039294 and GSK2315698
Description: as for outcome 25
Time Frame: as for outcome 32
Population: PK population. Data was not collected for Cohort 4a and 4b as study was terminated due to safety reasons during conduct of Part B (end of Cohort 3). Data was not calculated for Cohort 3 as the concentration-time data does not provide an accurate representation of the terminal elimination phase for the drug. Hence, AUC([0-inf]/D) was not derived.
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 0 | 0 | 0

35. Secondary Outcome: Part B: AUC(0-t) of GSK3039294 and GSK2315698
Description: as for outcome 26
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
h*ng/mL
  GSK3039294: Day 4 (n= 0, 0, 0): number analyzed (Participants) | 0 | 0 | 0
  GSK2315698: Day 4 (n= 7, 0, 0): number analyzed (Participants) | 7 | 0 | 0
  GSK2315698: Day 4 (n= 7, 0, 0) | 7571.9 (30.12) |  |
  GSK3039294: Day 5 (n= 0, 0, 0): number analyzed (Participants) | 0 | 0 | 0
  GSK2315698: Day 5 (n= 8, 0, 0) | 8900.1 (35.27) |  |

36. Secondary Outcome: Part B: AUC(0-t)/D of GSK3039294 and GSK2315698
Description: as for outcome 27
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL/mg
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
h*ng/mL/mg
  GSK3039294: Day 4 (n= 0, 0, 0): number analyzed (Participants) | 0 | 0 | 0
  GSK2315698: Day 4 (n= 7, 0, 0): number analyzed (Participants) | 7 | 0 | 0
  GSK2315698: Day 4 (n= 7, 0, 0) | 12.62 (30.12) |  |
  GSK3039294: Day 5 (n= 0, 0, 0): number analyzed (Participants) | 0 | 0 | 0
  GSK2315698: Day 5 (n= 8, 0, 0) | 14.83 (35.27) |  |

37. Secondary Outcome: Part B: Cmax of GSK3039294 and GSK2315698
Description: Blood samples were collected at specified time points for GSK3039294 and GSK2315698. Cmax was determined using standard non-compartmental methods. NA indicates data could not be calculated because only one participant was analyzed.
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
ng/mL
  GSK3039294: Day 4 (n= 3, 0, 0): number analyzed (Participants) | 3 | 0 | 0
  GSK3039294: Day 4 (n= 3, 0, 0) | 15.25 (55.24) |  |
  GSK2315698: Day 4 (n= 7, 0, 0): number analyzed (Participants) | 7 | 0 | 0
  GSK2315698: Day 4 (n= 7, 0, 0) | 1789.7 (29.75) |  |
  GSK3039294: Day 5 (n= 1, 0, 0): number analyzed (Participants) | 1 | 0 | 0
  GSK3039294: Day 5 (n= 1, 0, 0) | 16.70 (NA) — NA indicates data could not be calculated because only one participant was analyzed. |  |
  GSK2315698: Day 5 (n= 8, 0, 0) | 2652.6 (19.81) |  |

38. Secondary Outcome: Part B: Cmax/D of GSK3039294 and GSK2315698
Description: Blood samples were collected at specified time points for GSK3039294 and GSK2315698. Cmax/D was determined using standard non-compartmental methods. NA indicates that, data could not be calculated because only one participant was analyzed.
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
ng/mL/mg
  GSK3039294: Day 4 (n= 3, 0, 0): number analyzed (Participants) | 3 | 0 | 0
  GSK3039294: Day 4 (n= 3, 0, 0) | 0.025 (55.24) |  |
  GSK2315698: Day 4 (n= 7, 0, 0): number analyzed (Participants) | 7 | 0 | 0
  GSK2315698: Day 4 (n= 7, 0, 0) | 2.983 (29.75) |  |
  GSK3039294: Day 5 (n= 1, 0, 0): number analyzed (Participants) | 1 | 0 | 0
  GSK3039294: Day 5 (n= 1, 0, 0) | 0.028 (NA) — NA indicates that, data could not be calculated because only one participant was analyzed. |  |
  GSK2315698: Day 5 (n= 8, 0, 0) | 4.421 (19.81) |  |

39. Secondary Outcome: Part B: t1/2 of GSK3039294 and GSK2315698
Description: as for outcome 30
Time Frame: as for outcome 32
Population: PK population. Data was not collected for Cohort 4a and 4b as study was terminated due to safety reasons during conduct of Part B (end of Cohort 3). Data was not calculated for Cohort 3 as the concentration-time data does not provide an accurate representation of the terminal elimination phase for the drug. Hence, t1/2 was not derived.
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 0 | 0 | 0

40. Secondary Outcome: Part B: Tmax of GSK3039294 and GSK2315698
Description: as for outcome 31
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
Hours
  GSK3039294: Day 4 (n= 3, 0, 0): number analyzed (Participants) | 3 | 0 | 0
  GSK3039294: Day 4 (n= 3, 0, 0) | 0.500 [0.48 to 0.50] |  |
  GSK2315698: Day 4 (n= 7, 0, 0): number analyzed (Participants) | 7 | 0 | 0
  GSK2315698: Day 4 (n= 7, 0, 0) | 4.00 [4.00 to 5.95] |  |
  GSK3039294: Day 5 (n= 1, 0, 0): number analyzed (Participants) | 1 | 0 | 0
  GSK3039294: Day 5 (n= 1, 0, 0) | 0.500 [0.50 to 0.50] |  |
  GSK2315698: Day 5 (n= 8, 0, 0) | 6.00 [3.98 to 6.00] |  |

41. Secondary Outcome: Part B: Plasma Serum Amyloid P Component (SAP) Level of GSK3039294
Description: Blood samples were collected at specified time points for GSK3039294. Pharmacodynamic (PD) population consist of all participants who received at least one dose of study medication and who also had a baseline measurement and at least one post-treatment PD measure.
Time Frame: Cohort 3:Days1(pre-dose, 2hour post-dose),2(pre-dose),4(pre-dose),5(pre-dose, 30min,1,2,3,4,6 hours post-dose),7(pre-dose)and 21post-dose;Cohort4:Days1(pre-dose, 2 hour post-dose),2(pre-dose),4(pre-dose), 5(pre-dose, and 2 hours post-dose) and 35post-dose
Population: PD population. Data was not collected as study was terminated, due to safety reasons during conduct of Part B (end of Cohort 3) whereas Cohort 4a and 4b were not recruited in Part B. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294
Number analyzed (Participants) | 8 | 0 | 0
ng/mL
  Day 1: pre-dose (n=8, 0, 0) | 32318.69 (6403.13) |  |
  Day 1: 2 hour (n=8, 0, 0) | 4064.37 (761.37) |  |
  Day 2: pre-dose (n=8, 0, 0) | 939.83 (555.71) |  |
  Day 4: pre-dose (n=7, 0, 0): number analyzed (Participants) | 7 | 0 | 0
  Day 4: pre-dose (n=7, 0, 0) | 526.49 (303.64) |  |
  Day 5: pre-dose (n=8, 0, 0) | 456.28 (173.19) |  |
  Day 5: 30 min (n=7, 0, 0): number analyzed (Participants) | 7 | 0 | 0
  Day 5: 30 min (n=7, 0, 0) | 506.16 (232.88) |  |
  Day 5: 1 hour (n=8, 0, 0) | 458.72 (174.85) |  |
  Day 5: 2 hour (n=7, 0, 0): number analyzed (Participants) | 7 | 0 | 0
  Day 5: 2 hour (n=7, 0, 0) | 449.03 (160.56) |  |
  Day 5: 3 hour (n=8, 0, 0) | 366.31 (101.67) |  |
  Day 5: 4 hour (n=7, 0, 0): number analyzed (Participants) | 7 | 0 | 0
  Day 5: 4 hour (n=7, 0, 0) | 347.81 (115.59) |  |
  Day 5: 6 hour (n=8, 0, 0) | 264.79 (72.97) |  |
  Day 7: pre-dose (n=8, 0, 0) | 508.32 (301.64) |  |
  Day 21 (n=8, 0, 0) | 33320.64 (6252.46) |  |

42. Secondary Outcome: Part C: AUC(0-inf) of GSK3039294 and GSK2315698
Description: This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: Day 1 (pre-dose, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10 and 12 hours post-dose); Day 2 to 20 (pre-dose); Day 21 (pre-dose, and 0.5, 1, 2, 3, 4, 6, 8 and 12 hours post-dose; Week 4 and 5
Population: PK population. Data was not collected as study was terminated due to safety reasons during conduct of Part B (end of Cohort 3) whereas Part C was not initiated.
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

43. Secondary Outcome: Part C: AUC(0-inf)/D of GSK3039294 and GSK2315698
Description: This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: as for outcome 42
Population: as for outcome 42
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

44. Secondary Outcome: Part C: AUC(0-t) of GSK3039294 and GSK2315698
Description: This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: as for outcome 42
Population: as for outcome 42
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

45. Secondary Outcome: Part C: AUC(0-t)/D of GSK3039294 and GSK2315698
Description: This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: as for outcome 42
Population: as for outcome 42
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

46. Secondary Outcome: Part C: Cmax of GSK3039294 and GSK2315698
Description: This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: as for outcome 42
Population: as for outcome 42
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

47. Secondary Outcome: Part C: Cmax/D of GSK3039294 and GSK2315698
Description: This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: as for outcome 42
Population: as for outcome 42
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

48. Secondary Outcome: Part C: t1/2 of GSK3039294 and GSK2315698
Description: This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: as for outcome 42
Population: as for outcome 42
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

49. Secondary Outcome: Part C: Tmax of GSK3039294 and GSK2315698
Description: This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: as for outcome 42
Population: as for outcome 42
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

50. Secondary Outcome: Part C: Plasma SAP Levels of GSK3039294
Description: This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: as for outcome 42
Population: as for outcome 42
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

51. Secondary Outcome: Part C: Time to Repletion of SAP
Description: This analysis was planned but not performed for Part C as the study was terminated early during Part B.
Time Frame: as for outcome 42
Population: as for outcome 42
Arm/Group | Part C: GSK3039294
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Part A: Up to Day 14; Part B (Cohort 3: Up to Day 21, Cohort 4a and 4b: Up to Day 35); and Part C: Up to Day 63
Description: Safety population was analyzed which consisted of all participants who received at least one dose of the study medication. The study was terminated due to safety reasons during conduct of Part B (end of Cohort 3) whereas Cohort 4A and 4B were not recruited in Part B and Part C was not initiated.
Arm/Group | Part A: GSK3039294 200 mg | Part A: GSK3039294 600 mg | Part A: GSK3039294 1200 mg | Part B: Cohort 3- GSK3039294 600 mg QD | Part B: Cohort 4a- GSK3039294 | Part B: Cohort 4b- GSK3039294 | Part C: GSK3039294
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/16 | 0/8 | 0/8 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/16 | 0/8 | 1/8 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/8 | 6/16 | 5/8 | 7/8 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: GSK3039294 200 mg (N=8) | Part A: GSK3039294 600 mg (N=16) | Part A: GSK3039294 1200 mg (N=8) | Part B: Cohort 3- GSK3039294 600 mg QD (N=8) | Part B: Cohort 4a- GSK3039294 (N=0) | Part B: Cohort 4b- GSK3039294 (N=0) | Part C: GSK3039294 (N=0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: GSK3039294 200 mg (N=8) | Part A: GSK3039294 600 mg (N=16) | Part A: GSK3039294 1200 mg (N=8) | Part B: Cohort 3- GSK3039294 600 mg QD (N=8) | Part B: Cohort 4a- GSK3039294 (N=0) | Part B: Cohort 4b- GSK3039294 (N=0) | Part C: GSK3039294 (N=0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accelerated idioventricular rhythm (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT02603172/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT02603172/SAP_001.pdf